CLINICAL TRIAL: NCT05744882
Title: The Need Of Root Canal Treatment After Coronectomy In Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Rehan Ahmad, Rehan Ahmad, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIDM/ERC/12/2022/04
Record Dates: First submitted 2023-01-25; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Inferior Alveolar Nerve Injuries; Root Canal Treatment; Paresthesia; Third Molar; Impacted Third Molar Tooth; Coronectomy
MeSH Terms: conditions — Mandibular Nerve Injuries; Paresthesia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): no further treatment provided after coronectomy
  Interventions: Procedure: coronectony
- Experimental Group (Active Comparator): root canal treatment provided after the coronectomy procedure
  Interventions: Procedure: coronectony; Procedure: root canal treatment

INTERVENTIONS:
Procedure: coronectony — root canal treatment
  Other Names: procedure
Procedure: root canal treatment — root canal treatment
  Other Names: rct
  Arms: Experimental Group

SUMMARY:
The study included 24 patients with written and verbal consent Results with close proximity to IAN diagnosed based on radiographs and evaluation on the criteria of Howe, and Poyton were selected and divided into two groups by lottery method into coronectomy and coronectomy with root canal treatment following coronectomy groups. Patients were re-evaluated on three weeks for complications and three months follow-ups for radiographic evaluations of root-fragment migration

DETAILED DESCRIPTION:
The study enrolled 24 patients with written and verbal consent, out of which 15 were females and 9 were males aged between 18-30 years, with a mean age of males 24 ± 2.6 years and females 23.5 ± 2.8 years. Ethical approval was taken from the ethical review board of Altamash Institute of Dental Medicine with IRB No: AIDM/ERC/12/2022/04.

A total of 24 impacted mandibular teeth from 24 Patients with close proximity to IAN diagnosed based on radiographs and evaluation on the criteria of Howe and Poyton4 were selected for the purpose of this study. The timeline of the study was between January 2021 till January 2022.

The estimated sample size calculated for the study was 12 (6 participants in each group) which was raised to minimum of 24 (12 participants in each group). The calculations were performed using 12.5% as a proportion of infection in the control group and 87.5% as the proportion of infection in experimentation group from the study published by Sencimen et al.1 The software used for the sample size estimation was STATA 13.0 using "pearson's chi-squared test for two-samples proportions test". The following parameters were considered:

Alpha = 0.05 Power = 0.8 Delta = 0.75 Proportions of control group = 0.125 (12.5%) Proportions of Experimental group = 0.875 (87.5%) Considering the high lost to followup cases into account the sample size was raised to 24 participants with one tooth per individual. (ANNEXURE-I)

Patients were diagnosed and then referred to the Oral Maxillofacial department of Altamash Institute of Dental Medicine. Twenty-four patients with 24 impacted mandibular third molars were equally divided into a control group and a study group. Twelve patients in the study group had their root canal treatment after coronectomies while the other half, the control group only had their coronectomies done without any further procedure performed.

All the participants were equally divided into a control group and a study group by making them pick concealed envelopes containing a participant code for the participant allocation into groups. The experimental group contained twelve participants who had root canal treatment following coronectomies, while on the other hand, only coronectomies were performed in the rest of the participants without root canal treatment.

Patients who were willing and cooperative, along with no known uncontrolled medical conditions and no history of radiotherapy in the head and neck region, were included as a part of this research, while patients who showed resistance or were uncooperative, gave a history of uncontrolled medical condition, showed signs of local pathology or infection, history of radiotherapy in head and neck area were excluded from being included in the study.

All surgical procedures were performed under local anesthesia by the same surgeon. None of the patients were prescribed prophylactic antibiotics but were give a chlorhexidine mouth was a given before the procedure. Patients were prescribed post operative antibiotics with analgesics and thorough written instructions for proper wound care. A buccal approach for coronectomy was performed for all of them by the surgeon. Furthermore, all the endodontic treatment was performed by the same endodontist.

In the study group, the endodontist performed a pulpectomy and used a hypochlorite solution for irrigation of the canals. Finally, gutta-percha (GP) was used as a canal-filling material. All procedures performed by the endodontic followed the aseptic conditions and protocol.

The surgeon decided on a buccal approach with a three-cornered envelope incision resulting in a full thickness mucoperiosteal flap. The incision and eventually the flap was raised following the principles of incision and flap in order to promote a clean surgery leading to an uneventful and complication-free healing. The crown along the dental follicle was eliminated in addition to removing one-third of the root coronally.

The clinician decided on establishing a tilted or angled slope, the level of the slope descending lingually via buccal surface. This inclination resulted in a discrepancy of about 3-4mm in the levels of the corresponding root surfaces, consequence of which was a formation of a sharp edge on the buccal root surface. While the lingual root was 3-4mm below the lingual alveolar crest level. To compensate for the height, difference the buccal and lingual root surfaces, a reduction in the height of the buccal surface was performed in order to match with the lowered lingual root portion. Winding up the surgery with copious irrigation with saline followed by primary wound closure The mentioned step was carried out for both the study and the control group but in the in the study group, after removal of the pulp and biomechanical preparation, the canals were filled with GP. Multiple periapical radiographs were taken during endodontic procedure to ensure the correct filling of the canals and optimum filling till the apices.

More over the surgeon made a point to use a sharp bur for every operation in order to excise the crown without mobilizing the roots. In the control group the pulp was left in place. Follows up initially third week followed by sixth month were done with the help of panoramic radiograph.

ELIGIBILITY:
Inclusion Criteria:

* cooperative,
* no known uncontrolled medical conditions
* no history of radiotherapy in the head and neck region

Exclusion Criteria:

* not willing to participate
* history of uncontrolled medical condition
* sign of any local pathology
* history of radiotherapy in head and neck region

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Infection | 3 months
  Patients presenting with pain or swelling or both postoperatively within 3rd week to 3rd month of procedure. The the clinical presentation was confirmed by a clinician on clinical examination.

SECONDARY OUTCOMES:
Paresthesia | 3 months
  Patient presenting with history of numbness on any follow-up visit.
Movement of remnant root fragment | 3 months
  Apical movement remenant root fragment measured perpendicularly from occlusal plane by conparing pre-operative OPG-radiograph and another one taken at 3 month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Riordan BC. Coronectomy (intentional partial odontectomy of lower third molars). Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Sep;98(3):274-80. doi: 10.1016/S1079210404000496. PMID 15356463
- [Background] Renton T, Hankins M, Sproate C, McGurk M. A randomised controlled clinical trial to compare the incidence of injury to the inferior alveolar nerve as a result of coronectomy and removal of mandibular third molars. Br J Oral Maxillofac Surg. 2005 Feb;43(1):7-12. doi: 10.1016/j.bjoms.2004.09.002. PMID 15620767
- [Background] Howe, G.L. and Poyton, H.G. (1960) Prevention of Damage to the Inferior Dental Nerve during the Extraction of Mandibular Third Molars. British Dental Journal, 109, 355-363.
- [Background] MERRILL RG. DECOMPRESSION FOR INFERIOR ALVEOLAR NERVE INJURY. J Oral Surg Anesth Hosp Dent Serv. 1964 Jul;22:291-300. No abstract available. PMID 14155469
- [Background] Kubota S, Imai T, Nakazawa M, Uzawa N. Risk stratification against inferior alveolar nerve injury after lower third molar extraction by scoring on cone-beam computed tomography image. Odontology. 2020 Jan;108(1):124-132. doi: 10.1007/s10266-019-00438-2. Epub 2019 Jun 17. PMID 31209581
- [Background] Cilasun U, Yildirim T, Guzeldemir E, Pektas ZO. Coronectomy in patients with high risk of inferior alveolar nerve injury diagnosed by computed tomography. J Oral Maxillofac Surg. 2011 Jun;69(6):1557-61. doi: 10.1016/j.joms.2010.10.026. Epub 2011 Feb 1. PMID 21288616
- [Background] Monaco G, D'Ambrosio M, De Santis G, Vignudelli E, Gatto MRA, Corinaldesi G. Coronectomy: A Surgical Option for Impacted Third Molars in Close Proximity to the Inferior Alveolar Nerve-A 5-Year Follow-Up Study. J Oral Maxillofac Surg. 2019 Jun;77(6):1116-1124. doi: 10.1016/j.joms.2018.12.017. Epub 2018 Dec 31. PMID 30689961
- [Background] Leung YY, Cheung LK. Long-term morbidities of coronectomy on lower third molar. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Jan;121(1):5-11. doi: 10.1016/j.oooo.2015.07.012. Epub 2015 Jul 22. PMID 26337212
- [Background] Pedersen MH, Bak J, Matzen LH, Hartlev J, Bindslev J, Schou S, Norholt SE. Coronectomy of mandibular third molars: a clinical and radiological study of 231 cases with a mean follow-up period of 5.7years. Int J Oral Maxillofac Surg. 2018 Dec;47(12):1596-1603. doi: 10.1016/j.ijom.2018.06.006. Epub 2018 Jul 14. PMID 30017572
- [Background] Dalle Carbonare M, Zavattini A, Duncan M, Williams M, Moody A. Injury to the inferior alveolar and lingual nerves in successful and failed coronectomies: systematic review. Br J Oral Maxillofac Surg. 2017 Nov;55(9):892-898. doi: 10.1016/j.bjoms.2017.09.006. Epub 2017 Oct 20. PMID 29061470
- [Background] Nishimoto RN, Moshman AT, Dodson TB, Beirne OR. Why Is Mandibular Third Molar Coronectomy Successful Without Concurrent Root Canal Treatment? J Oral Maxillofac Surg. 2020 Nov;78(11):1886-1891. doi: 10.1016/j.joms.2020.05.046. Epub 2020 Jun 11. PMID 32640205
- [Background] Valmaseda-Castellon E, Berini-Aytes L, Gay-Escoda C. Inferior alveolar nerve damage after lower third molar surgical extraction: a prospective study of 1117 surgical extractions. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Oct;92(4):377-83. doi: 10.1067/moe.2001.118284. PMID 11598570
- [Background] Pitros P, Jackson I, O'Connor N. Coronectomy: a retrospective outcome study. Oral Maxillofac Surg. 2019 Dec;23(4):453-458. doi: 10.1007/s10006-019-00794-x. Epub 2019 Aug 27. PMID 31456131
- [Background] Frenkel B, Givol N, Shoshani Y. Coronectomy of the mandibular third molar: a retrospective study of 185 procedures and the decision to repeat the coronectomy in cases of failure. J Oral Maxillofac Surg. 2015 Apr;73(4):587-94. doi: 10.1016/j.joms.2014.10.011. Epub 2014 Oct 22. PMID 25544301
- [Background] Kohara K, Kurita K, Kuroiwa Y, Goto S, Umemura E. Usefulness of mandibular third molar coronectomy assessed through clinical evaluation over three years of follow-up. Int J Oral Maxillofac Surg. 2015 Feb;44(2):259-66. doi: 10.1016/j.ijom.2014.10.003. Epub 2014 Nov 8. PMID 25457826
- [Background] Patel V, Sproat C, Kwok J, Beneng K, Thavaraj S, McGurk M. Histological evaluation of mandibular third molar roots retrieved after coronectomy. Br J Oral Maxillofac Surg. 2014 May;52(5):415-9. doi: 10.1016/j.bjoms.2014.02.016. Epub 2014 Mar 29. PMID 24684971
- [Result] Sencimen M, Ortakoglu K, Aydin C, Aydintug YS, Ozyigit A, Ozen T, Gunaydin Y. Is endodontic treatment necessary during coronectomy procedure? J Oral Maxillofac Surg. 2010 Oct;68(10):2385-90. doi: 10.1016/j.joms.2010.02.024. Epub 2010 Jul 21. PMID 20663600